CLINICAL TRIAL: NCT02766491
Title: Improving Stretching Interventions for Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Barbara Kalkman, Principal Investigator, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Stretching_CP_V1
Record Dates: First submitted 2016-04-19; First posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Cerebral Palsy
Keywords: Stretching
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strengthening and stretching (Experimental): The intervention group will follow a strengthening-stretching program of the calf muscles.
  Interventions: Other: Strengthening and stretching
- conventional stretching (Active Comparator): The control group will receive conventional stretching and strengthening exercises to the upper limb to assure that the same systemic physiological stimuli and a similar number of contact hours is received.
  Interventions: Other: conventional stretching

INTERVENTIONS:
Other: Strengthening and stretching — Strengthening exercises will be performed 4 times a week for 10 weeks. Single leg heel raises will be the preferred exercise performed. The group of participants will have a wide range of strength and functional abilities, this will be accounted for with individualised programmes. The exercise load can be reduced by switching to bilateral heel raises, giving external support, reducing the range of motion or performing the heel raises while seated. Exercise load will be progressively increased by adding weight in the form of water bottles to a rucksack worn on the participant's back.
  For the final six weeks of the intervention, stretching exercises of the calf muscles will be performed.
  Arms: Strengthening and stretching
Other: conventional stretching — This group will perform seated biceps curls 4 times a week for 10 weeks, where extra load can be added progressively by holding water bottles in the hand.
  For the final six weeks of the intervention, stretching exercises of the calf muscles will be performed.
  Arms: conventional stretching

SUMMARY:
Cerebral palsy (CP) has a prevalence of 1.5-3 per 1000 live births, making it the most common neurological disorder among children in Europe. One of the most frequently observed problems in CP is hypertonia, i.e. increased muscle tension, which can result in contractures. Stretching therapies are widely used as a treatment for contractures, but with highly variable success. Therefore, efforts are needed to improve the efficacy of stretching interventions. The investigators hypothesise that increasing the stiffness of the tendon relative to the muscle, by resistance training, prior to stretching will improve the efficacy of stretching interventions in children with CP. In a RCT design the investigators will compare a group of children receiving a combined strengthening-stretching intervention of the calf muscle to a control group receiving conventional stretching exercises in combination with upper limb exercises. Outcome measures will include muscle-tendon structure and gait analysis to assess functional improvements. This research will improve the understanding of muscle responses to stretching interventions in children with CP and can lead to more effective stretching therapies.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a disorder resulting from a non-progressive lesion in the brain during pregnancy or early childhood. Children with CP show impaired movement patterns compared to typically developing (TD) children. One of the main factors limiting movement in children with CP is a reduced range of motion (ROM), which can be caused by a combination of neural and mechanical factors. Mechanical factors contributing to a reduced ROM are increased muscle/fascicle stiffness, reduced muscle length and changes in intramuscular tissue properties, all of which contribute to contractures.

Contractures are conservatively treated with stretching therapies, e.g., casting, night splints and physical therapy. However, they are very demanding for both children and parents, especially physical therapy which is painful and time-consuming. Therefore, when recommending stretching therapies, we need to assure they are efficacious. However, recent reviews show that the outcomes of stretching therapies in children with CP are highly variable.

Stretching interventions aim to improve ROM motion by increasing the overall length and/or lengthening properties of the muscle. To successfully achieve these adaptations, the muscle must experience adequate tensile stimulus during the intervention. However, it has been shown by previous studies examining muscle behaviour during stretch, that the muscle and fascicles in children with CP lengthen less than in TD children. Our own studies have confirmed this observations at the muscle, but also shown that the tendon in children with CP lengthens more during a stretch, than in TD children. These observations indicate that the higher stiffness of the target muscle relative to the in series tendon prevents the muscle fibres to experience a sufficiently large stretching stimulus, and the adaptations are small. Accordingly, in a recent study on long term stretching interventions it has been shown that muscle and fascicle strain increase, but no changes in the muscle's resting length or functional improvements have been found.

If you were to increase the stiffness of the tendon relative to the muscle prior to the stretching intervention, a greater stretching stimulus could be provided to the muscle. This would mean that for any given joint stretch the muscle will experience a greater portion of the stretch. It is well established in healthy adults and children that the stiffness of the tendon increases following resistance training. Given that well-designed resistance training is effective and safe for children with CP, the same increased tendon stiffness should follow gains in muscle strength in this group too. It is therefore hypothesise that a combined strengthening-stretching intervention would stiffen the tendon, increase the amount of stretch seen by the muscle, and thereby improve the effectiveness of stretching interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with spastic cerebral palsy
* GMFCS level I-III
* Have the ability to perform at least one bi-lateral heel raise.
* Aged 7 to 14

Exclusion Criteria:

* Orthopaedic or neural surgery to the lower limb 2 years prior to or planned during the intervention
* Botulinum Toxin A injections 6 months prior to or planned during the intervention.
* A learning or behaviour impairment that prevents full participation in the intervention.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change Muscle fascicle length of the Gastrocnemius (mm) | at baseline and after 10 weeks
  B-mode ultrasound images will be captured at the mid muscle belly. From these, fascicle length will be defined as the straight line distance between the upper and the lower aponeurosis parallel to the lines of collagenous tissue.
Change in Gastrocnemius muscle length (mm) | at baseline and after 10 weeks
  B-mode ultrasound images will be captured of the myotendinous junction and the medial femoral condyl. Muscle length will be defined as the straight line distance between these two anatomical points.

SECONDARY OUTCOMES:
Change in ankle range of motion (degree) | at baseline and after 10 weeks
  The difference in ankle angle measured at maximal plantar flexion and maximal dorsi flexion with a goniometer
Change in Achilles tendon stiffness (Nm) | at baseline, after 4 weeks and after 10 weeks
  Tendon stiffness is quantified as the change in tendon length per change in tendon force. Tendon lengthening will be quantified, using B-mode ultrasound, from the displacement of the myotendinous junction during the MVC trials.
  Tendon force will be calculated from the ratio of nett joint moment to Achilles tendon moment arm.
Change in maximal dorsiflexion angle during gait (degree) | at baseline and after 10 weeks
  Maximal dorsiflexion angles will be quantified from kinematic data obtained during the gait analysis
Change in lengthening properties of the muscle fascicles (mm) | at baseline and after 10 weeks
  The ankle will be moved passively through the full range of motion. B-mode ultrasound images of the mid belly of the medial gastrocnemius will be collected throughout on which muscle fascicle lengthening will be measured
Changes in step length during gait (m) | at baseline and after 10 weeks
  Step length will be quantified from the kinematic data obtained during the gait analysis
Changes in ankle power at push of during gait | at baseline and after 10 weeks
  Ankle power will be quantified from kinematic and kinetic data obtained during the gait analysis

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D O'Brien, PhD, Study Director — Liverpool John Moores University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalkman BM, Holmes G, Bar-On L, Maganaris CN, Barton GJ, Bass A, Wright DM, Walton R, O'Brien TD. Resistance Training Combined With Stretching Increases Tendon Stiffness and Is More Effective Than Stretching Alone in Children With Cerebral Palsy: A Randomized Controlled Trial. Front Pediatr. 2019 Aug 13;7:333. doi: 10.3389/fped.2019.00333. eCollection 2019. PMID 31456995